CLINICAL TRIAL: NCT01815229
Title: Sore Throat Secondary to Endotracheal Intubation: the Role of Neutrophil Activation
Brief Title: Role of Neutrophil Activation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 201301037
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Results first posted 2019-07-15 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-05

CONDITIONS: Patients Requiring Endotracheal Intubation
Keywords: endotracheal; intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- tracheal lavages (Experimental): After the placement of the endotracheal tube (Hi-Lo™ Evac Mallinckrodt), tracheal lavages will be performed.
  A simultaneous blood sample of approx 5cc, will be collected by venipuncture or by sampling from intravenous or arterial line if available. The same procedure for collection of tracheal sample and blood will be repeated at the end of the surgical procedure and immediately prior to removal of the ETT. A total of approx 10cc blood will be collected for research purposes.
  Interventions: Procedure: tracheal lavages
- Healthy Control (Placebo Comparator): To replicate activation, neutrophils were isolated from 30mL blood of healthy volunteers and cocultured with TLF from subjects with or without sore throat pain.
  Interventions: Procedure: tracheal lavages

INTERVENTIONS:
Procedure: tracheal lavages — tracheal lavages obtained during endotracheal intubation.

SUMMARY:
Patients will undergo placement of an endotracheal tube (ETT) as standard of care. Tracheal lavage will be conducted using 5 mL of sterile saline solution by a push/suction technique. Specimen samples obtained by wall suction will be collected at 2 time points following intubation.

Blood samples will be obtained at 2 time points, simultaneous with the collection of the tracheal specimens.

ELIGIBILITY:
Inclusion Criteria

1. Ages 18 to 65
2. American Society of Anesthesiologists Physical Status Classification (ASA) I and II
3. Required to have endotracheal intubation
4. Scheduled for short admission (<23 hrs), or ambulatory orthopedic surgery (ankle, shoulder, or extremity surgery); general surgery (exploratory laparotomy, cholecystectomy, ventral or inguinal hernia repair); obstetric/gynecological surgery(total abdominal hysterectomy, bilateral salpingo-oophorectomy); urologic surgery (nephrectomy, prostatectomy), lumbar spine surgery( discectomy, one or two level lumbar fusion) procedures.
5. Estimated duration of surgery 3 to 4 hours.
6. Provide informed consent

Exclusion Criteria

1. Active pulmonary disease within 5 days prior to enrollment
2. On immunosuppressive medications
3. Previous tracheal surgery
4. On azithromycin
5. Diabetes
6. Pregnancy
7. Smoking history of less than 6 weeks prior to surgery
8. Surgery or intubation within 5 days of surgery
9. Planned surgical procedure involving neck or thoracic regions
10. Active pulmonary disease
11. Autoimmune disease (HIV, AIDS, Rheumatoid Arthritis
12. Hepatitis
13. Cancer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-03; Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Puyo, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Tracheal Lavages Sore Throat; Tracheal Lavages No Sore Throat: After the placement of the endotracheal tube (Hi-Lo™ Evac Mallinckrodt), tracheal lavages will be performed.
  A simultaneous blood sample of approx 5cc, will be collected by venipuncture or by sampling from intravenous or arterial line if available. The same procedure for collection of tracheal sample and blood will be repeated at the end of the surgical procedure and immediately prior to removal of the ETT. A total of approx 10cc blood will be collected for research purposes.
  tracheal lavages: tracheal lavages obtained during endotracheal intubation.
- Healthy Control: A one time blood sample of approx 30cc will be collected by venipuncture.
Period: Overall Study
Arm/Group | Tracheal Lavages Sore Throat | Tracheal Lavages No Sore Throat | Healthy Control
Started | 13 | 18 | 51
Completed | 13 | 18 | 0
Not Completed | 0 | 0 | 51

BASELINE CHARACTERISTICS:
Groups:
- Tracheal Lavages No Sore Throat: After the placement of the endotracheal tube (Hi-Lo™ Evac Mallinckrodt), tracheal lavages will be performed.
  A simultaneous blood sample of approx 5cc, will be collected by venipuncture or by sampling from intravenous or arterial line if available. The same procedure for collection of tracheal sample and blood will be repeated at the end of the surgical procedure and immediately prior to removal of the ETT. A total of approx 10cc blood will be collected for research purposes.
- Healthy Control: To replicate activation, neutrophils were isolated from 20mL blood of healthy volunteers and cocultured with TLF from subjects with or without sore throat pain.
- Total: Total of all reporting groups
Arm/Group | Tracheal Lavages Sore Throat | Tracheal Lavages No Sore Throat | Healthy Control | Total
Number analyzed (Participants) | 13 | 18 | 51 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 18 | 51 | 82
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] — Population: Age collected categorically for healthy controls. Unable to calculate mean values.
  years
    age /years: number analyzed (Participants) | 13 | 18 | 0 | 31
    age /years | 40.92 [26 to 56] | 40.78 [19 to 61] |  | 41.17 [19 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Sex: Female | 8 | 7 | 31 | 46
  Sex: Male | 5 | 11 | 20 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 6 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 5 | 16 | 23
  White | 9 | 13 | 29 | 51
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 13 | 18 | 51 | 82

OUTCOME MEASURES:

1. Primary Outcome: Neutrophil Cell Counts in Tracheal Lavages
Description: Neutrophil cell count were collected after an average of 3.2 hours of exposure to an ETT. Cell counts were performed using 10x6 per ml
Time Frame: average of 3.2 hours of exposure to an ETT
Population: Blood samples were collected form healthy controls for in vitro analysis. Neutrophil data was not collected for healthy controls.
Measure: Mean (Standard Deviation); unit: neutrophil/high powered field
Groups:
- Tracheal Lavage no Sore Throat: After the placement of the endotracheal tube (Hi-Lo™ Evac Mallinckrodt), tracheal lavages will be performed.
  A simultaneous blood sample of approx 5cc, will be collected by venipuncture or by sampling from intravenous or arterial line if available. The same procedure for collection of tracheal sample and blood will be repeated at the end of the surgical procedure and immediately prior to removal of the ETT. A total of approx 10cc blood will be collected for research purposes.
  tracheal lavages: tracheal lavages obtained during endotracheal intubation.
Arm/Group | Tracheal Lavages Sore Throat | Tracheal Lavage no Sore Throat
Number analyzed (Participants) | 13 | 18
neutrophil/high powered field
  IL-1β | 112.02 (150.53) | 26.98 (59.42)
  TNF-α | 61.72 (72.64) | 27.63 (34.99)
  Il-8 | 6513.22 (5209.84) | 1995.59 (2262.19)
Statistical Analysis 1: Comparison: Tracheal Lavages Sore Throat vs Tracheal Lavage no Sore Throat; Tracheal lavages (TL) were done in intubated humans to obtain cell counts; Test type: Other; p < 0.05, t-test, 2 sided — P value applies to cell count at removal

2. Secondary Outcome: Intubation Time in Minutes
Description: Average amount of time that participants were intubated
Time Frame: Up to 363 minutes for intubation time
Population: Healthy control were not intubated.
Measure: Mean (Full Range); unit: minutes
Arm/Group | Tracheal Lavages Sore Throat | Tracheal Lavage no Sore Throat
Number analyzed (Participants) | 13 | 18
minutes | 213 [123 to 354] | 175 [55 to 363]

ADVERSE EVENTS:
Time Frame: approximately 5 hours per participant
Arm/Group | Tracheal Lavages Sore Throat | Tracheal Lavages No Sore Throat | Healthy Control
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/18 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/18 | 0/51
Other Adverse Events (participants affected / at risk) | 0/13 | 0/18 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-11): https://cdn.clinicaltrials.gov/large-docs/29/NCT01815229/Prot_SAP_000.pdf